CLINICAL TRIAL: NCT02560571
Title: Preoperative Evaluation of Endometrial Cancer
Brief Title: Pre-operative Studies for Prediction of Lymph Nodes Involvement in Endometrial Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Yfat kadan, Dr, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0142-15-MMC
Record Dates: First submitted 2015-09-21; First posted 2015-09-25 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Ultrasonography; Hematologic Tests

ARMS (1):
- all patients (Experimental): all study patients will undergo ultrasound and blood test
  Interventions: Device: ultrasound; Other: blood test

INTERVENTIONS:
Device: ultrasound
Other: blood test

SUMMARY:
The study evaluates pre-operative prediction of the risk for lymph nodes involvement in endometrial cancer patients. Patients will undergo ultrasound exam (bi and three dimensional) and biomarker test - Ca 125, in addition to routine physical and laboratory exams, before surgery.

The sonographic evaluation will include endometrial characteristics and myometrial invasion, pelvic findings and enlarged lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial cancer patients
* Surgical candidates

Exclusion Criteria:

* Fertility preservation therapy
* Contraindication for surgery
* Stage 2 and higher

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
number of participants with positive nodes | 4 weeks after surgery (4-6 weeks from enrollment)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center, Kfar Saba, Israel